CLINICAL TRIAL: NCT02162121
Title: Stimulating Catheter for Lumbar Plexus Block: Better Postoperative Analgesia?
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: ASST Gaetano Pini-CTO (Other)
Responsible Party: Principal Investigator, Gianluca Cappelleri, Medical Doctor, ASST Gaetano Pini-CTO
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IOGPGC06-14
Record Dates: First submitted 2014-06-09; First posted 2014-06-12 (Estimated); Last update posted 2017-08-14 (Actual); Status verified 2017-08

CONDITIONS: Hip Replacement Arthroplasty
MeSH Terms: interventions — Anesthesia, Spinal; Ketorolac

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stimulating catheter (Experimental): After Spinal Anesthesia (Levobupivacaine 0,5% 15mg) all patients in the arm will receive continuous lumbar plexus block with stimulating catheter ("Stimolong", "Pajunk", Germany). Mepivacaine 1% 15 ml will be administrated. As post-operative analgesia Ropivacaine 0,2% will be continuous administrated.
  Interventions: Procedure: Continuous lumbar plexus: stimulating catheter; Procedure: Spinal Anesthesia; Procedure: Local anesthetic infusion; Procedure: Intravenous analgesia; Procedure: Opioids rescue analgesia; Drug: Mepivacaine 1%; Drug: Levobupivacaine 0,5%; Drug: Ropivacaine 0,2%; Drug: Ketorolac 30mg; Drug: Buprenorphine 0,2mg; Device: Stimulong, Pajunk, Germany.
- Non-stimulating catheter (Active Comparator): After Spinal Anesthesia (levobupivacaine 0,5% 15mg) all patients in the arm will receive continuous lumbar plexus block with non-stimulating catheter ("Stimolong", "Pajunk", Germany). Mepivacaine 1% 15ml will be administrated. As post-operative analgesia Ropivacaine 0,2% will be continuous administrated.
  Interventions: Procedure: Spinal Anesthesia; Procedure: Local anesthetic infusion; Procedure: Intravenous analgesia; Procedure: Opioids rescue analgesia; Drug: Mepivacaine 1%; Drug: Levobupivacaine 0,5%; Drug: Ropivacaine 0,2%; Drug: Ketorolac 30mg; Drug: Buprenorphine 0,2mg; Device: Stimulong, Pajunk, Germany.; Procedure: Continuous lumbar plexus: non-stimulating catheter

INTERVENTIONS:
Procedure: Continuous lumbar plexus: stimulating catheter — Perinervous stimulating catheter ("Stimulong", "Pajunk", Germany) will be insert in lumbar plexus through tuohy needle (18G, 100mm length). 15ml mepivacaine 1% are injected before the complete resolution of the spinal anesthesia.
  Arms: Stimulating catheter
Procedure: Spinal Anesthesia — Spinal anesthesia will be perform at L3-L4 or L4-L5 level. Levobupivacaine 0,5% 15mg will be injected.
Procedure: Local anesthetic infusion — Continuous infusion (Mini Rythmic Evolution, Micrel) of ropivacaine 0,2% at 3ml/h, bolus 3 ml, lockout time 15 min, 12 ml/h maximum dose through perinervous catheter until 3rd postoperative day
Procedure: Intravenous analgesia — Ketorolac 30mg 3 times a day
Procedure: Opioids rescue analgesia — Buprenorphine 0,2mg twice a day if VAS>4
Drug: Mepivacaine 1%
Drug: Levobupivacaine 0,5%
Drug: Ropivacaine 0,2%
Drug: Ketorolac 30mg
Drug: Buprenorphine 0,2mg
Device: Stimulong, Pajunk, Germany.
Procedure: Continuous lumbar plexus: non-stimulating catheter
  Arms: Non-stimulating catheter

SUMMARY:
Stimulating catheters have been introduced to reduce the incidence of secondary failure after continuous peripheral nerve blocks, but they effectiveness over traditional nonstimulating catheters is still controversial. The aim of this prospective, randomized, blinded study is to detect if stimulating catheters improve postoperative compared with conventional non-stimulating catheters.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing total hip arthroplasty

Exclusion Criteria:

* diabetes neurological disorders coagulation disorders rheumatoid arthritis chronic opioids therapy allergy to local anesthetic

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2014-05; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Local anesthetic consumption | 72h
  Evaluation of local anesthesic consumption every 6h in first 72 postoperative hours.

SECONDARY OUTCOMES:
Visual Analog scale (VAS) score | 72h postoperatively
  Evaluation of VAS static and VAS dynamic during first 72 postoperative hours
Up and Go test | 4th postoperative day
  "up and go" test: time need to get up from a chair, walk for 3 meters, and come back to seat down on the chair
Opioids request | 72h postoperatively
  Opioids consumption will be recorded throughout 72 postoperative hours
Quadriceps strength | preoperative and 24h, 48h, 72h postoperatively
  evaluate bilateral muscle strength with an isometric force dynamometer to measure the force produced during a maximum voluntary isometric contraction in a lying position by the knee flex to 90°.
postoperative nausea and vomiting (PONV) | 72h postoperatively
  Evaluation of nausea and vomit incidence in postoperative period with scale 0 from 4
Needle redirections | During catheter position
  During catheter positioning number of needle redirections necessary to found lumbar plexus are recorder.
Catheter insertion time | During catheter positioning
  Time (minutes) needed for catheter placement

CONTACTS AND LOCATIONS:
Overall Officials: Gianluca Cappelleri, M.D., Principal Investigator — ASST Gaetano Pini-CTO
Locations (1):
- Istituto ortopedico Gaetano Pini, Milan, Italy